CLINICAL TRIAL: NCT01847651
Title: LOLA in Hepatic Encephalopathy Brain Muscle Axis During Treatment of Hepatic Encephalopathy With L-ornithine L-aspartate A Phase iv Randomised Double Blind Placebo- Controlled Trial
Brief Title: Brain Muscle Axis During Treatment of Hepatic Encephalopathy With L-ornithine L-aspartate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOLA-Merz WMDH P39937; 2012-003817-32 (EudraCT Number); 12/LO/1937 (Other: Research Ethics Committee (REC)); CRO2033 (Other: Imperial College London Reference)
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2013-05

CONDITIONS: Hepatic Encephalopathy; Minimal Hepatic Encephalopathy; Cirrhosis
Keywords: hepatic encephalopathy; minimal hepatic encephalopathy; cirrhosis; lateral vastus; muscle biopsy; L ornithine L aspartate; functional magnetic resonance imaging; magnetic resonance spectroscopy; cognitive testing; Paper and pencil Hepatic Encephalopathy score (PHES); Cogstate; urine metabonomics; plasma metabonomics; muscle metabonomics
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Blood Specimen Collection; Nutrition Assessment; Spectrum Analysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOLA (Active Comparator): Other Names:
  Hepa-Merz Granulat 3000 Hepa-Merz granules 3g (Each 5g sachet contains 3g of L-ornithine L-aspartate) L-ornithine L-aspartate LOLA
  Randomised to a daily dose 18g per day, two sachets of Hepa-Merz granules three times a day (or placebo)
  Interventions: Procedure: Vastus Muscle Biopsy; Drug: LOLA or placebo; Other: Cognitive assessment (PHES); Other: Cognitive Assessement (Cogstate); Other: blood and urine sampling; Other: Nutritional assessment; Other: MRI brain and spectroscopy; Other: MRI leg cross section; Other: Functional MRI (working memory and attention tasks)
- Placebo (Placebo Comparator)
  Interventions: Procedure: Vastus Muscle Biopsy; Drug: LOLA or placebo; Other: Cognitive assessment (PHES); Other: Cognitive Assessement (Cogstate); Other: blood and urine sampling; Other: Nutritional assessment; Other: MRI brain and spectroscopy; Other: MRI leg cross section; Other: Functional MRI (working memory and attention tasks)

INTERVENTIONS:
Procedure: Vastus Muscle Biopsy — Both Arms, all 3 visits at 0, 4 and 12 weeks
Drug: LOLA or placebo — Hepa-Merz Granulat 3000 Hepa-Merz granules 3g (Each 5g sachet contains 3g of L-ornithine L-aspartate) L-ornithine L-aspartate LOLA Randomised to a daily dose 18g per day, two sachets of Hepa-Merz granules three times a day (or placebo)for 12 weeks
Other: Cognitive assessment (PHES) — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: Cognitive Assessement (Cogstate) — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: blood and urine sampling — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: Nutritional assessment — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: MRI brain and spectroscopy — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: MRI leg cross section — Both Arms, all 3 visits at 0, 4 and 12 weeks
Other: Functional MRI (working memory and attention tasks) — Both Arms, all 3 visits at 0, 4 and 12 weeks

SUMMARY:
Patients with cirrhosis of the liver may suffer from a condition called hepatic encephalopathy which in its mildest form as mental slowing and impaired reaction times in driving and machinery operation. Left untreated it may lead to deep coma. The cause is not fully understood but is though to be related to the inability of a damaged liver to filter out toxins such as ammonia in the blood, which then accumulate within the brain and result in altered function and swelling within certain brain cells,astrocytes. These patients also suffer from muscle loss, which is associated with a poor outcome. L-ornithine L-aspartate(LOLA) is a licensed drug in Germany and has been shown to promote ammonia elimination from the body in the form of urea. Some experimental studies have suggested that LOLA also potentially attenuates muscle loss by incorporating ammonia into muscle in the form of glutamine. The aim of this study is to determine cognitive and nutritional effects of 12 weeks of LOLA administration and its effect on brain muscle structure and function in patients with cirrhosis.

DETAILED DESCRIPTION:
This is a Phase IV randomised double blind, placebo controlled study. Thirty four patients with cirrhosis will be studied with psychometric tests, clinical brain magnetic resonance imaging(MRI),including functional MRI) and magnetic resonance spectroscopy (MRS) and muscle MRI of leg muscle before (time 0)during (4weeks)and after LOLA or placebo treatment at 12 weeks. Samples will also be taken for ex vivo MRS of blood and urine to identify potential biomarkers. Histological analysis and MRS would also be performed on the muscle tissue at the same time points.

Hypotheses Primary objective

1) Improvement in mental state by paper and pencil based Psychometric Hepatic Encephalopathy Score (PHES) and Cogstate Research test (computer based cognitive research assessment tool)

Secondary objectives

1. Brain volume reduction due to reduction in brain swelling measured by MRI and improvement in the chemical structure of the brain due to (cerebral osmolytes)measured by in vivo MR Spectroscopy (MRS)scanning of the brain.
2. Improvement in brain function
3. Improvement in muscle function (muscle metabolome normalisation) and increased muscle size (fat free mass), measured in vivo by MRI scanning and by in vitro mass spectroscopy and NMR spectroscopy and histological analysis of muscle samples.
4. Improvement in the chemical profile of key chemicals in the blood and urine, measured with in vitro NMR spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* Ambulant patients of any Child-Pugh stage cirrhosi and PHEs defined MHe or grade 1 encephalopathy

Exclusion Criteria:

* Previous episodes of overt HE without a clear precipitant
* Recurrent excessive alcohol consumption (abstinence for those with alcoholic liver disease otherwise less than 28 units per week)
* Severe coagulopathy (INR>2, platelets <60 000/uL, Fibrinogen <1mg/dl)
* known myopathy or myositis, taruma to lower extremities within 3 months)
* Renal dysfunction with a serum creatinine>3mg/dl (265micromol/L)
* Ferromagnetic implants
* Recent intestinal haemorrhage within 1 month
* Claustrophobia
* Weight >120kg
* Major psychoactive medication such as antipsychotic agents
* Known cerebrovascular disease or pre-existing neurological conditions
* Age less than 18 or greater than 65.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Improvement in mental state on paper and pencil Hepatic Encephalopathy score (PHES) testing and Cogstate testing (computer based cognitive assessment research tool) | At 0, 4 and 12 weeks

SECONDARY OUTCOMES:
Brain Volume | At 0 , 4 and 12 weeks
  The effect of brain volume reduction due to reduction of brain swelling will be measured by serial brain MRI (at 0, 4 and 12 weeks)
Brain chemical structure | 0, 4, 12 weeks
  Improvement in brain chemical structure (by measuring cerebral osmolytes) will be assessed by in-vivo MR spectroscopy
Improvement in brain function measured by functional MRI | 0, 4, 12 weeks
  Key brain functions such as attention and working memory (the default mode network) will be assessed through fMRI
Improvement in Muscle Function and increase in muscle size | 0, 4 and 12 weeks
  Increase in muscle size(fat free mass) will be measured on by MR imaging of the thigh, in-vitro NMR spectroscopy, mass spectroscopy and histological analysis of muscle biopsy samples.
Improvement of plasma and urine metabolome | 0, 4 and 12 weeks
  Improvement in blood and urine profiles will be measured with in vitro NMR spectroscopy to assess for biomarkers of treatment response and to determine the amino acids altered by treatment of HE.

CONTACTS AND LOCATIONS:
Overall Officials: Simon D Taylor-Robinson, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Liver unit St Mary's Hospital, 10th floor QEQM Wing, South Wharf Road, London, London, United Kingdom